CLINICAL TRIAL: NCT05451628
Title: Anatomy-Based Fitting in Unexperienced Cochlear Implant Users
Acronym: ABFmulti
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Universitair Ziekenhuis Brussel (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: EC-2021-437
Record Dates: First submitted 2022-06-02; First posted 2022-07-11 (Actual); Last update posted 2023-12-12 (Actual); Status verified 2023-12

CONDITIONS: Cochlear Implants; Sensorineural Hearing Loss
MeSH Terms: conditions — Hearing Loss, Sensorineural

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Default CI fitting (Active Comparator): Programming of cochlear implant speech processor according to standard clinical care
  Interventions: Device: Default CI fitting
- Anatomy-based CI fitting (Active Comparator): Programming of cochlear implant speech processor with anatomy-based fitting
  Interventions: Device: Anatomy-based CI fitting

INTERVENTIONS:
Device: Default CI fitting — Programming of cochlear implant speech processor according to standard clinical care
  Arms: Default CI fitting
Device: Anatomy-based CI fitting — Programming of cochlear implant speech processor with anatomy-based fitting
  Arms: Anatomy-based CI fitting

SUMMARY:
Severe to profound hearing loss affects 0,8% of the global population. For these people, a conventional hearing aid often does not provide sufficient benefit. However, these people can benefit from a cochlear implant (CI). A CI needs to be individually programmed (fitted) for each recipient. A fitting "map" is defined as a set of electrical parameters that are individually adapted to a recipient's needs to achieve optimal sound perception. At present, most CI recipients are fitted with a default frequency allocation map that doesn't take individual variability in size and shape of the cochlea into account. In this study, a fitting strategy based on the post-operative CT scan, that will allow the audiologist to set a frequency-band distribution for CI fitting that may be more closely aligned to the natural tonotopic frequency distribution of a normal hearing cochlea, will be evaluated.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years
* Post-lingual onset of severe to profound sensory-neural hearing loss in the implanted ear(s)
* Post-operative Computed Tomography (CT) scan of the CI electrode available
* Pre-operative result of pure-tone audiometry, speech test in quiet and in noise available
* Subject implanted with MED-EL cochlear implant(s)
* Subjects received a Flex28, FlexSoft or Standard electrode
* Subject planned to receive a SONNET 2 or RONDO 3 audio processor on the newly implanted side
* Audio processor not yet activated on the newly implanted side
* The most apical active electrode contact has to be inserted at least 450°
* Minimum of 10 active channels can be activated
* Fluent in the language of the test centre
* Signed and dated Informed Consent Form (ICF) before the start of any study-specific procedure

Exclusion Criteria:

* Lack of compliance with any inclusion criteria
* Electric Acoustic Stimulation (EAS) user (user of an EAS audio processor)
* Implanted with C40+, C40X and C40C
* Implanted with an Auditory Brainstem Implant (ABI) or Split electrode array
* Anything that, in the opinion of the Investigator, would place the subject at increased risk or pre-clude the subject's full compliance with or completion of the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2022-03-30 (Actual); Primary Completion 2025-01 (Estimated); Study Completion 2025-01 (Estimated)

PRIMARY OUTCOMES:
Speech recognition test in quiet (S0): percentage correctly identified phonemes | 3 months post-activation
Speech recognition test in quiet (S0): percentage correctly identified phonemes | 6 months post-activation

SECONDARY OUTCOMES:
Speech recognition test in noise (S0N0): the speech reception threshold in dB SNR | 3 months post-activation
Speech recognition test in noise (S0N0): the speech reception threshold in dB SNR | 6 months post-activation
Result of the pitch matching test: frequency difference in semitones | 3 months post-activation
Result of the pitch matching test: frequency differences in semitones | 6 months post-activation
Result of the perception of timbre test: Score on Visual Analog Scale (VAS) | 3 months post-activation
  Patients have to rate the timbre on a visual analog scale (VAS) ranging from 0 to 10, where a higher score reflects a better outcome.
Result of the perception of timbre test: Score on Visual Analog Scale (VAS) | 6 months post-activation
  Patients have to rate the timbre on a visual analog scale (VAS) ranging from 0 to 10, where a higher score reflects a better outcome.
Result of the consonance and dissonance rating test: Plot of pleasantness over frequency interval and modulation measure | 3 months post-activation
Result of the consonance and dissonance rating test: Plot of pleasantness over frequency interval and modulation measure | 6 months post-activation
Result of the speech contrast discrimination test: Psychometric function of phoneme categorization | 3 months post-activation
Result of the speech contrast discrimination test: Psychometric function of phoneme categorization | 6 months post-activation
Patient reported outcome- Hearing Implant Sound Quality Index (HISQUI): Total score and classification of self-perceived auditory benefit | 1 day visit (At the activation of the sound processor)
Patient reported outcome- Hearing Implant Sound Quality Index (HISQUI): Total score and classification of self-perceived auditory benefit | 3 months post-activation
Patient reported outcome- Hearing Implant Sound Quality Index (HISQUI): Total score and classification of self-perceived auditory benefit | 6 months post-activation
Datalogging data: Average numbers of hours per day | 2 weeks post-activation
Datalogging data: Average numbers of hours per day | 1 months post-activation
Datalogging data: Average numbers of hours per day | 3 months post-activation
Datalogging data: Average numbers of hours per day | 6 months post-activation

CONTACTS AND LOCATIONS:
Overall Officials: Vedat Topsakal, Prof., Principal Investigator — UZB-VUB
Locations (1):
- UZ Brussel, Brussels, Belgium

IPD SHARING:
Plan to Share IPD: No